CLINICAL TRIAL: NCT06971328
Title: Effects of Acceptance and Commitment-Based (ACT) Psychoeducation on Caregiver Burden, Posttraumatic Growth and Psychological Resilience in Caregivers of Patients With Schizophrenia
Brief Title: ACT-Based Psychoeducation for Schizophrenia Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Merve Bakar Gürcüoğlu, Nursing, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-MBG-01
Record Dates: First submitted 2025-04-15; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia Patients

STUDY DESIGN:
Intervention Model Description: In order to prevent bias in the study, the pre-test, post-test and follow-up application will be conducted by the interviewer. Data from the experimental and control groups will be collected simultaneously. Individuals in both groups will be interviewed one-on-one, and the psychoeducation application will be applied individually to the experimental group. Written and verbal consent will be obtained from the caregivers, and an explanation will be made regarding the purpose of the study. The Sociodemographic Data Form, Zarit Caregiver Burden, Post-Traumatic Development, and Brief Psychological Resilience Scale (Appendix 1) created by the researcher at the beginning of the study will be applied to the control group, and the control group, which received the pre-test, will be monitored. No application will be made to the control group. Afterwards, the forms specified in the pre-test will be applied to the control group, which will be monitored for 8 weeks, as a post-test. A follow-up test
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: • During the data evaluation process, the data of the experimental and control groups will be given a code (random, from 1 to 34) to ensure blinding of the statistician. In this way, the triple blinding method will be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deney Grubu (Experimental): ACT-based psychoeducation will be applied to schizophrenia caregivers in the experimental group.
  Interventions: Other: ACT-based psychoeducation
- Kontrol grubu (No Intervention): Schizophrenia caregivers in the control group will be monitored without any intervention.

INTERVENTIONS:
Other: ACT-based psychoeducation — It is thought that ACT-based psychoeducation will be an effective psychiatric nursing practice in reducing the care burden of individuals caring for schizophrenia patients and increasing their post-traumatic development and psychological resilience. However, no study has been found in the literature evaluating the effects of these three parameters. In general, the number of ACT-based psychoeducation studies applied to schizophrenia caregivers is quite low. Three thesis studies were found in our country, and no study examining the effect of ACT-based psychoeducation on the post-traumatic development levels of schizophrenia caregivers was found in the domestic and foreign literature. Based on this gap in the literature, the planned study is aimed to be presented to the literature as an intervention that can be used in holistic psychiatric nursing care and to reveal its effects in the specified parameters.
  Arms: Deney Grubu

SUMMARY:
Schizophrenia is an important mental health problem that requires caregivers because it causes disability. With the efforts to move from a hospital-based model to a community-based model in mental health services, the care of schizophrenia patients is mainly provided by their families at home, creating a significant care burden on caregivers or, on the contrary, post-traumatic development is reported. Psychiatric nurses are responsible for evaluating the patient together with their family by taking these conditions into consideration when providing care to individuals with mental illness. As a principle of humanistic and holistic care, nursing interventions to be implemented by psychiatric nurses to develop caregivers' coping methods, reduce their care burden and contribute to their post-traumatic development are extremely important in terms of the effectiveness and efficiency of care. Acceptance and Commitment (ACT)-based psychoeducation, whose effectiveness has been reported in the literature, is an important application in providing care to patients and families in psychiatric nursing practices. ACT is among the third generation therapies that aim to keep individuals in the moment with awareness, adopt the willingness to accept events instead of struggling with them, and create an important source of power in taking actions in line with life values. In this study, 17 out of 34 individuals determined by statistical methods among the caregivers of schizophrenia patients will be included in the control group and monitored, while 17 will receive 8 sessions of ACT-based psychoeducation in the intervention group, and the effects of the education on caregiver burden, post-traumatic development, and psychological resilience will be evaluated. There are very few studies in the literature where ACT-based psychoeducation is applied to caregivers of schizophrenia patients. Although studies examining the effects on individuals' caregiver burden and psychological resilience are limited, no study has been found examining its effects on post-traumatic development, and this constitutes the original value of the study. As a result of this study, it is expected that ACT-based education will reduce the caregiver burden in schizophrenia caregivers and increase their psychological resilience through post-traumatic development.

DETAILED DESCRIPTION:
Schizophrenia is a significant mental health problem in terms of its prevalence and disability. Individuals who experience significant loss of professional/social functioning and inability to perform self-care activities need a caregiver. Many physical, psychological, and economic problems and a related high care burden have been reported in caregivers. These difficulties increase the entry of caregivers into the health system along with sick individuals, contributing to the increase in health costs and mental problems. Studies have shown that interventions to be applied to caregivers will reduce the care burden and increase the coping capacities of individuals. While a relative being diagnosed with schizophrenia can cause trauma in individuals in itself, on the contrary, they can also experience post-traumatic development, and their high post-traumatic development is effective in reducing the care burden experienced by caregivers. Another important factor in caregivers' struggle with the mentioned difficulties is psychological resilience. Interventions to strengthen psychological resilience are gaining importance in this context. Considering the contemporary roles of psychiatric nursing, it is inevitable for the family to be treated holistically, to reduce the burden of care, and to provide therapeutic interventions that will strengthen the caregiver spiritually. When the literature is examined, it is seen that Acceptance and Commitment (ACT) based interventions are highly effective for individuals providing care to schizophrenia patients, but it is noteworthy that there are not enough studies. In particular, no study has been found examining the effect of ACT based psychoeducation on the post-traumatic development levels of caregivers. This study was planned to reveal the effect of Acceptance and Commitment based psychoeducation applied to individuals providing care to schizophrenia patients on the burden of care, post-traumatic development, and psychological resilience of individuals in order to contribute to its inclusion in psychiatric nursing practices.

ELIGIBILITY:
Inclusion Criteria:

* Providing primary care to an individual diagnosed with schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) V
* Living with the patient and providing care for at least 6 months
* Being over 18 years of age
* Being literate
* Not having been diagnosed with any mental illness
* Agreeing to participate in the study and being a volunteer

Exclusion Criteria:

* The patient must live in a different house and spend less than 6 hours together per day
* Having previously attended ACT or Psychoeducation programs

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Data Form | The measurement tests to be applied to the experimental and control groups will be the first test at the beginning of the study, the second test 8 weeks after the beginning, and the follow-up test four weeks after the second test.
  The experimental and control groups will be given a pre-test at the beginning of the study, a post-test after 8 weeks, and a follow-up test after four weeks. The questionnaire form to be applied in the pre-test and post-test is the Sociodemographic Data Form prepared by the researcher. Sociodemographic Data Form prepared by the researcher. The sociodemographic data form consists of age, gender, marital status, education level, degree of closeness to the patient, and duration of care.

SECONDARY OUTCOMES:
Zarit Caregiver Burden Scale | The measurement tests to be applied to the experimental and control groups will be the first test at the beginning of the study, the second test 8 weeks after the beginning, and the follow-up test four weeks after the second test.
  Zarit Caregiver Burden Scale (scale consists of 19 items and will be scored from 1 to 5 from low to high (never, rarely, occasionally, quite often, almost always).

OTHER OUTCOMES:
Posttraumatic Growth Questionnaire | The measurement tests to be applied to the experimental and control groups will be the first test at the beginning of the study, the second test 8 weeks after the beginning, and the follow-up test four weeks after the second test.
  The other scale used is the 21-item Posttraumatic Growth Questionnaire (scale from 0 to 5; never experienced, very little experienced, somewhat experienced, moderately experienced, very experienced, very experienced)
Brief Resilience Scale | The measurement tests to be applied to the experimental and control groups will be the first test at the beginning of the study, the second test 8 weeks after the beginning, and the follow-up test four weeks after the second test.
  Another scale used is the 6-item Brief Resilience Scale (scoring from low to high; not at all appropriate, not appropriate, somewhat appropriate, appropriate, completely appropriate)

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Şehir Hastanesi, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No